CLINICAL TRIAL: NCT00372970
Title: Randomized Placebo-Controlled Double Blind Study of Botulinum Toxin Versus Placebo for the Treatment of Gastroparesis
Brief Title: Placebo Controlled Trial of Botulinum Toxin for Gastroparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Principal Investigator, Frank K. Friedenberg, Professor of Medicine, Temple University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4204
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-05

CONDITIONS: Gastroparesis
Keywords: gastroparesis; vomiting; nausea; bloating; dyspepsia
MeSH Terms: conditions — Gastroparesis; Vomiting; Nausea; Dyspepsia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin A (Active Comparator): 200 U of Botox injected endoscopically into pylorus
  Interventions: Drug: Botulinum toxin A
- Placebo (Placebo Comparator): saline into pylorus.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum toxin A — 200 U given by injection into the pylorus.
  Other Names: Botox into pylorus
  Arms: Botulinum Toxin A
Drug: Placebo — saline injection into pylorus.
  Other Names: saline injection into pylorus
  Arms: Placebo

SUMMARY:
It is hypothesized that in some patients with gastroparesis increased pyloric tone may be a contributing feature. Botox relaxes the pylorus so that food can empty the stomach more rapidly. Lesser quality studies have shown that this treatment works in about 40% of patients, and relieves symptoms for up to 3 months. This study compares this treatment to placebo (saline) injection. After a 1 month period patients may elect to receive open label botox who have not received relief from their first injection. Patients symptoms and gastric emptying are followed for 1 year.

DETAILED DESCRIPTION:
Patients with gastroparesis, or delayed gastric emptying, present with early satiety, postprandial bloating, nausea, vomiting, and abdominal pain or discomfort.1 Gastric emptying is a highly regulated process reflecting the integration of propulsive forces generated by proximal fundic tone and distal antral contractions with the resistance of the pyloric sphincter. Antral hypomotility as well as increased gastric outlet resistance due to pyloric dysfunction or pylorospasm appear to be important physiologic disturbances in gastroparesis.2-4 Current treatment for gastroparesis employs prokinetic agents that increase antral contractility and accelerate gastric emptying.5 Unfortunately, prokinetic agents have limited efficacy and trials of these agents have suffered from significant methodological flaws.6 Troublesome side effects such as cardiac arrhythmias in the case of cisapride (Propulsid, Janssen Pharmaceutica) and extrapyramidal symptoms and sedation in the case of metoclopramide (Reglan, A.H. Robins) have limited the usefulness of these agents.7 Domperidone may be effective for treating symptoms of gastroparesis, however it is unavailable in the U.S.8

Botulinum toxin (Botox, Allergan) is an inhibitor of cholinergic neuromuscular transmission and has been used to treat spastic disorders of both striated and smooth muscles by local injection into affected muscles.9 Previous published work from our institution demonstrated that injection of botulinum toxin into the pylorus improved gastric emptying and reduces symptoms in idiopathic gastroparesis.10 In our open label study, patients had a 38% reduction in gastroparesis symptoms when interviewed 4 weeks after injection. Seventy percent of patients had improved gastric emptying. No immediate or short term (within 6 months) untoward events occurred in our study. The beneficial effect of botulinum toxin injection was suggested to be through decreasing pyloric resistance; however, manometric analysis of this region was not performed. Our results are similar to those seen in other studies that have demonstrated accelerated gastric emptying in response to pyloric botulinum toxin injection.11-13 These studies have included groups of patients with both idiopathic and diabetic gastroparesis. Unfortunately, in all studies, the patient groups have been very small and the study design has been open label that might bias results in favor of a positive response. In addition, follow-up has been for only 6 months.

Despite limited data, many gastroenterologists are now using botulinum toxin injection for the treatment of gastroparesis outside the context of clinical research studies. We are concerned that this practice may be increasing nationwide without definitive proof of efficacy. A randomized, placebo-controlled trial is necessary to establish the usefulness of pyloric botulinum toxin injection for gastroparesis. Botulinum toxin therapy is expensive and may not be efficacious. In addition, if efficacious, the mechanism by which botulinum toxin improves gastric emptying needs to be studied. This research protocol will answer several questions concerning this potentially useful therapy for gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Documented gastroparesis by radiologic study
* No ulcer disease
* Only surgery history must be either appendectomy or cholecystectomy
* No prior treatment with Botox

Exclusion Criteria:

* Prior botox injection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank K Friedenberg, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Friedenberg FK, Palit A, Parkman HP, Hanlon A, Nelson DB. Botulinum toxin A for the treatment of delayed gastric emptying. Am J Gastroenterol. 2008 Feb;103(2):416-23. doi: 10.1111/j.1572-0241.2007.01676.x. Epub 2007 Dec 5. PMID 18070232

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients all recruited at Temple University Hospital from 7/1/2005 to 9/1/2007
Groups:
- Botulinum Toxin: Received 200U of Botox injected into pyloric sphincter endoscopically.
- Placebo: Received 5 cc saline injected into pyloric sphincter endoscopically.
Period: Overall Study
Arm/Group | Botulinum Toxin | Placebo
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients with documented gastroparesis
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (11.6) | 40.4 (13.0) | 41.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Symptom Response as Assessed by the Gastroparesis Cardinal Symptom Index.
Description: Scale for GI symptoms related to gastroparesis. For this we will use the gastroparesis cardinal symptom index (GCSI).
  The GCSI is based on three subscales: post-prandial fullness/early satiety (4 items); nausea/vomiting (3 items), and bloating (2 items). Scores range from 0-5 for the nine items and an asymptomatic patient would have a score of 0 with a highly symptomatic patient having a score of 45. For this study the score had to be >=27. In a previous study internal consistency reliability was 0.84 for the GCSI total score and ranged from 0.83 to 0.85 for the subscale scores. Two week test retest reliability was 0.76 for the total score and ranged from 0.68 to 0.81 for subscale scores.
Time Frame: 1 month
Population: All patients had gastroparesis and underwent EGD. Injection double blinded.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Botox: Botox injection into pylorus
Arm/Group | Botox | Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 6.8 (9.2) | 10.1 (12.7)

ADVERSE EVENTS:
Arm/Group | Botox | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 6/16 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botox (N=16) | Placebo (N=16)
Headache (Nervous system disorders) | 6 (6) | 3 (3)
Fatigue (Nervous system disorders) | 3 (3) | 3 (3)
Other (General disorders) | 0 (0) | 0 (0) — Not serious adverse event
other (General disorders) | 0 (0) | 0 (0) — other non-serious events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No